CLINICAL TRIAL: NCT00213252
Title: Can Montelukast Shorten Corticosteroid Therapy In Children With Mild To Moderate Acute Asthma?
Brief Title: Use of Montelukast to Treat Children With Mild to Moderate Acute Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Merck Frosst Canada Ltd. (Industry)
Responsible Party: Principal Investigator, Suzanne Schuh, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1000007674
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Asthma, Bronchial
Keywords: asthma, randomized trial, pediatrics
MeSH Terms: conditions — Asthma | interventions — montelukast; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Montelukast plus prednisolone
- 2 (Active Comparator)
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Montelukast plus prednisolone — Single dose of oral prednisolone with a subsequent daily five-day course of oral Montelukast
  Arms: 1
Drug: Prednisolone — Six daily doses of oral prednisolone
  Arms: 2

SUMMARY:
The primary objective of this study is to evaluate if children with acute asthma given a single dose of oral prednisolone with a subsequent daily five-day course of oral Montelukast will achieve a therapeutic failure rate at day 8 not significantly higher than those given six daily doses of oral prednisolone. Secondary objectives include comparison of the two groups with respect to the changes in symptoms, beta2 agonists, clinical asthma score and days without asthma by day 8.

DETAILED DESCRIPTION:
We plan a randomized double blind double-dummy trial of 190 previously healthy children 2-17 years of age presenting to the Emergency Department (ED) at the Hospital for Sick Children in Toronto with mild to moderate acute asthma, with the Pulmonary Index score ≤ 11 points and PRAM ≤ 8 points. Asthma will be defined as at least the second episode of wheezing, with signs of lower airway obstruction. All participating children will receive a single dose of oral prednisolone 2mg/kg (max 60 mg) on arrival and standardized inhaled salbutamol in the ED and for five days thereafter. At discharge from ED children will be randomized to two interventional groups. Those in the Montelukast group will get oral Montelukast 4 mg (2-5 year olds), 5 mg (6-14 year olds), and 10 mg (15-17 year olds) as well as daily prednis(ol)one placebo 24 hours after the ED dose of prednisolone and at 48, 72, 96 and 120 hours, while those in the prednisolone group will receive Montelukast placebo and daily oral prednisolone 1mg/kg (max 60 mg) for five further doses at these times.

The primary outcome will be therapeutic failure in the two groups from randomization to day 8. This failure will be defined as unscheduled medical visits for asthma symptoms or hospitalization or treatment with oral corticosteroids outside the experimental protocol. Secondary outcome measures include comparison of the number of salbutamol treatments, changes in the previously validated daytime symptoms scale, nighttime cough/awakening scale, number of asthma-free days within the 8 day observational period in the two groups, changes in the PI and PRAM scores to 48 hours and day 8 as well as the association between the main treatment effect and age, pulmonary index at randomization and history of atopy.

This study will take two 9 months periods. Primary analysis will include a one-sided 95% CI for the difference in failure rate in the prednisolone group minus the Montelukast group. Secondary analyses will include repeated measures ANOVA for differences in changes of continuous variables and the Fisher's Exact test for comparison of proportions. An exploratory sub-group logistic regression analysis will be done for examining interaction between the main treatment effect and possible covariates.

In the event that the patients given a single dose of prednisolone followed by Montelukast have comparable therapeutic failure rate to those given standard extended prednisolone therapy, administration of Montelukast may help us abbreviate the length of corticosteroid therapy in children with acute asthma.

ELIGIBILITY:
Inclusion Criteria:

* age 2-17 years
* Clinical diagnosis of mild to moderate asthma as a second wheezing episode associated with signs of respiratory distress suggesting lower airway obstruction such as tachypnea and/or use of accessory muscles of respiration.
* baseline Pulmonary Index Clinical Score (Appendix B) ≤ 11 out of 15 possible points as well as PRAM ≤ 8 out of 12 points.
* Presenting to the Sick Kids Emergency Department
* Children capable of FEV1 measurement will have FEV1 more than 60% of the predicted value
* male or female
* Willing and able to provide informed consent (or informed consent by parents)

Exclusion Criteria:

* No previous history of wheezing or bronchodilator therapy. This population may eventually have diagnoses other than asthma or viral induced wheezing
* Patients who received more than a single dose of oral corticosteroids within 72 hours prior to arrival
* Patients receiving more than 500 mcg per day of fluticasone for more than 1 month or more than 250 mcg of fluticasone for more than 7 days prior to arrival
* Patients who have had more than 2 previous visits to the asthma clinic at SickKids
* Patients who received Montelukast within one week of arrival
* Critically ill patients requiring airway stabilization
* Patients with severe asthma, defined as PI 12 to 15 or PRAM 9 to 12.
* Co-existent co-morbidities such as chronic pulmonary disease and cardiac disease requiring pharmacotherapy, neurologic disease and immune disorders.
* Previous admission to ICU for asthma.
* More than 3 hospitalizations for asthma during the past 12 months.
* Contact with varicella within the previous 21 days.
* Insufficient command of the English language

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2005-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Therapeutic failure rate | From randomization at discharge from the Emergency Department to day 8

SECONDARY OUTCOMES:
Number of inhaled salbutamol treatments | From randomization to 24, 48, 72, 96, 120, 144 hours and day 8
Change in the daytime asthma symptom scale from randomization | 48 hours and Day 8
Change in the nighttime cough | 8 days
Number of days without asthma | 8 days
Change in the Pulmonary Index Score from baseline | 48 hours and Day 8
Change in the Pediatric Respiratory Assessment Measure(PRAM)from baseline | 48 hours and Day 8
Association between the main treatment effect and patients' age, disease severity at randomization (Pulmonary Index and PRAM) and personal/family history of atopy. | 48 hours and Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Schuh, MD, Principal Investigator — The Hospital for Sick Children, Toronto, Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Result] Schuh S, Willan AR, Stephens D, Dick PT, Coates A. Can montelukast shorten prednisolone therapy in children with mild to moderate acute asthma? A randomized controlled trial. J Pediatr. 2009 Dec;155(6):795-800. doi: 10.1016/j.jpeds.2009.06.008. Epub 2009 Aug 4. PMID 19656525